CLINICAL TRIAL: NCT00804310
Title: Phase I Study of Lapatinib (GW572016) in Combination With Weekly Ixabepilone (BMS 247550) in Advanced Solid Tumors
Brief Title: Lapatinib and Ixabepilone in Treating Patients With Advanced Solid Tumors
Acronym: UCDCC#207
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000626165; P30CA093373 (NIH)
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — ixabepilone; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lapatinib and Ixabepilone (Experimental)
  Interventions: Drug: ixabepilone; Drug: lapatinib ditosylate

INTERVENTIONS:
Drug: ixabepilone — This intravenous treatment will be performed on an outpatient basis. Ixabepilone (15 - 20mg/m2) will be given weekly for 3 weeks, then one week off, every 28 days (4 weeks). The study doctor will decide how long to keep the participant on this treatment based on how the participant is tolerating the drug and how it is affecting the tumor.
  Other Names: Ixempra
Drug: lapatinib ditosylate — Lapatinib (1000-1500 mg) will be administered orally on a daily basis. The study doctor will decide how long to keep the participant on this treatment based on how the participant is tolerating the drug and how it is affecting the tumor.
  Other Names: Tykerb/Tyverb

SUMMARY:
RATIONALE: Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as ixabepilone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving lapatinib together with ixabepilone may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of lapatinib given together with ixabepilone in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the safety and feasibility of lapatinib ditosylate in combination with ixabepilone in patients with advanced solid tumors.

Secondary

* To determine the maximum-tolerated dose of this regimen in these patients.
* To assess, preliminarily, the efficacy of this regimen in these patients.
* To perform laboratory correlative studies on tissue and blood specimens from these patients to investigate potential predictors of response.

OUTLINE: This is a multicenter, dose-escalation study.

Patients receive oral lapatinib ditosylate once daily on days 1-28 and ixabepilone IV on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Archival tumor tissue samples are collected for EGFR/HER2 pathway analyses via immunohistochemistry, mRNA analysis via RT-PCR, EGFR mutation analyses, Kras and braf mutation analysis via sequencing, and RAS mutations via PCR and sequencing. Blood samples are also collected periodically for tumor DNA and proteomics, acetylated alpha-tubulin analysis, EGFR-HER2 pathway genotypes, and pharmacogenomics.

After completion of study therapy, patients are followed for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have cytologically or histologically proven advanced solid tumors for which there is no known standard therapy available or are not eligible for standard therapy because of their performance status, or have progressed after standard therapy.
* Patients must have measurable or evaluable disease
* Patients must be 18 years of age or older
* Patients must have a Zubrod performance status of 0-2
* Patients must have an estimated survival of at least 3 months
* Any prior chemotherapy must have been completed at least 3 weeks prior to start of this protocol and all side effects (except alopecia) resolved to grade 1 or less. Any prior radiation must have been completed at least 2 weeks prior to start of therapy. Patients must have completed prior trastuzumab (Herceptin) at least 4 weeks prior to start of protocol therapy
* Patients must have adequate renal function
* Patients must have adequate liver function
* Patients must have a pretreatment granulocyte count of >1500/mm3 and platelet count of >100 000/mm3.
* Patients must have a cardiac ejection fraction within the institutional range of normal as measured by 2-D echocardiogram or MUGA scan.
* All patients must give informed consent
* Patients must be able to take and retain oral medication
* Patients of reproductive potential must agree to use an effective contraceptive method while on treatment as the effects of these drugs on the unborn fetus are unknown.

Exclusion Criteria:

* Patients may not have previously received lapatinib, ixabepilone or any other EGFR-TKI targeted agent. Prior trastuzumab (Herceptin) is allowed.
* Patients may not pregnant or breastfeeding as the effects of these drugs on the unborn fetus are unknown.
* Patients with symptomatic brain metastasis or still requiring steroids and anticonvulsants may not participate. Patients with asymptomatic treated brain metastasis (surgical resection or radiotherapy) may be included if they are neurologically stable and have been off steroids for at least 2 weeks.
* Patients with pre-existing neuropathy > grade 2 may not participate.
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, will be excluded.
* History of other diseases, metabolic dysfunction, physical examination finding or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the patient at high risk from treatment complications.
* Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, or prior surgical procedures affecting absorption.
* HIV-positive patients receiving combination antiretroviral therapy are excluded from the study because of possible pharmacokinetic interactions with lapatinib. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Patients requiring oral anticoagulants are eligible provided there is appropriate close INR monitoring in place.
* Prior radiation must not have included more than 30% of bone marrow containing areas
* Any prior, severe history of hypersensitivity reaction to a drug formulated in CremaphorEL
* Adherence to the requirements for concomitant medications classified as CYP3A4 inducers or inhibitors, or gastric pH modifiers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-08; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Safety and Toxicity | Toxicity will be assessed at the beginning of every cycle and on day 8 and 15 of every cycle for at least eight weeks (2 cycles). Maximum of 6 cycles.
  Assessed by NCI CTCAE v 3.0

SECONDARY OUTCOMES:
Maximum tolerated dose (MTD) | One cycle (4 weeks)
Preliminary efficacy | One year

CONTACTS AND LOCATIONS:
Overall Officials: Helen K. Chew, MD, Principal Investigator — University of California, Davis
Locations (4):
- United States (4):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana